CLINICAL TRIAL: NCT01959100
Title: Evaluation of the Efficacy of Azithromycin to Prevent Bronchiolitis Obliterans Syndrome After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy of Azithromycin to Prevent Bronchiolitis Obliterans Syndrome After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ALLOZITHRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P120110
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Malignant Hematological Diseases
Keywords: hematopoietic stem cell transplantation; pulmonary non-infectious complications; bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycine (Experimental): 250 mg x 3/week during a meal for a period of 2 years
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): 250 mg x 3/week during a meal for a period of 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — 250 mg x 3/week per os during a meal for a period of 2 years
  Arms: Azithromycine
Drug: Placebo — 250 mg x 3/week during a meal for a period of 2 years
  Arms: Placebo

SUMMARY:
The occurrence of bronchiolitis obliterans syndrome (SBO) after allogeneic hematopoietic stem cell transplantation (HSCT) is considered to be a chronic pulmonary graft versus host disease (GVHD) that is associated with significant mortality and morbidity. The reported incidence of SBO varies from 6 to 26% of allogeneic HSC recipients and is usually diagnosed within 2 years after transplantation. The diagnosis of SBO relies on the occurrence of a new airflow obstruction identified during pulmonary function testing, and the definition differs between studies. Currently, no curative immunosuppressive treatment is available, and recent data suggest that the use of these treatments, especially corticosteroids, should be limited because of their toxicity. The impairment of lung function parameters is likely caused by fibrous small airway lesions. Few data on the pathogenesis of SBO after allogeneic HSCT are available. Several hypotheses are based on the occurrence of SBO during chronic graft rejection after lung transplantation, which shares many clinical and histopathological similarities with SBO after allogeneic HSCT. One hypothesis is that the first step leading to SBO is lung epithelium injury. SBO is then identified as an alloimmune reaction with only one clearly identified risk factor: extrathoracic chronic GVHD. Due to their anti-inflammatory and immunomodulatory properties, recent data suggest that low-dose macrolides may be effective at preventing SBO after lung transplants. This well-tolerated treatment may be useful for preventing SBO after allogeneic HSCT.

The objective of this Phase 3 multicentre randomized, double-blinded, clinical trial is to evaluate the efficacy of azithromycin in preventing BO syndrome after allogeneic HSCT in patients with malignant hematological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 16 years old
* Experimenting an allogeneic HSCT for a hematologic malignancy
* Pre-transplantation Pulmonary Function Testing
* With written informed consent

Exclusion Criteria:

* Allergy or Intolerance to azithromycin, macrolides or ketolide or excipient
* Prolonged corrected QT (QTc) interval (>450 msec)
* Taking medications that prolong the QTc interval (Cisapride, ergotamine, dyhydroergotamine)
* Taking ergotamine and dyhydroergotamine due to the risk of ergotism
* Family history of a prolonged QTc interval.
* History of congestive heart failure
* Taking colchicine Severe liver insufficiency • History of infection due to atypical mycobacteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Airflow decline (AFD)-free survival | 2 year after allogeneic HSCT
  Defined on the criteria from Chien JW et al (Am J Resp Crit Care Med 2003;168:208-14) by an annualized decline of percent predicted forced expiratory volume in 1 second (FEV1) of more than 5%

SECONDARY OUTCOMES:
Overall survival | within 2 years of inclusion
Occurrence of late-onset pulmonary non-infectious complications (=bronchiolitis obliterans syndrome, SBO) | within 2 years after inclusion
  bronchiolitis obliterans syndrome (SBO) is defined as the absence of infection with an forced expiratory volume in 1 second (FEV1) of <75% of predicted or a decline of > 10% and FEV1/Slow vital capacity (SVC) < 0.7 or residual volume (RV) or RV/total lung capacity (TLC) > 120%, and interstitial lung disease, which is defined as the onset of new interstitial lung abnormalities observed with a lung CT scan and the absence of infection.
Variation of pulmonary function testing parameters | within 2 years after inclusion
  variation in mean forced expiratory volume in 1 second (FEV1) decline, forced vital capacity (FVC), residual volume (RV), Total Lung capacity (TLC), Forced expiratory flow at 25% point to the 75% point of Forced Vital Capacity (FEF25-75%) as compared to baseline values (at inclusion)
Occurrence of acute and chronic extra-thoracic graft versus host disease (GVHD) | within 2 years after inclusion
Cumulative incidence of hematological relapse | within the 2 years after inclusion
Quality of life | within 2 years after inclusion
Tolerance | within 2 years of inclusion
  adverse events
Cumulative dose of steroids treatment | within the 2 years after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Bergeron A, Chevret S, Chagnon K, Godet C, Bergot E, Peffault de Latour R, Dominique S, de Revel T, Juvin K, Maillard N, Reman O, Contentin N, Robin M, Buzyn A, Socie G, Tazi A. Budesonide/Formoterol for bronchiolitis obliterans after hematopoietic stem cell transplantation. Am J Respir Crit Care Med. 2015 Jun 1;191(11):1242-9. doi: 10.1164/rccm.201410-1818OC. PMID 25835160
- [Derived] Vallet N, Le Grand S, Bondeelle L, Hoareau B, Corneau A, Bouteiller D, Tournier S, Derivry L, Bohineust A, Tourret M, Gibert D, Mayeur E, Itzykson R, Pacchiardi K, Ingram B, Cassonnet S, Lepage P, Peffault de Latour R, Socie G, Bergeron A, Michonneau D. Azithromycin promotes relapse by disrupting immune and metabolic networks after allogeneic stem cell transplantation. Blood. 2022 Dec 8;140(23):2500-2513. doi: 10.1182/blood.2022016926. PMID 35984904
- [Derived] Bergeron A, Chevret S, Granata A, Chevallier P, Vincent L, Huynh A, Tabrizi R, Labussiere-Wallet H, Bernard M, Chantepie S, Bay JO, Thiebaut-Bertrand A, Thepot S, Contentin N, Fornecker LM, Maillard N, Risso K, Berceanu A, Blaise D, Peffault de La Tour R, Chien JW, Coiteux V, Socie G; ALLOZITHRO Study Investigators. Effect of Azithromycin on Airflow Decline-Free Survival After Allogeneic Hematopoietic Stem Cell Transplant: The ALLOZITHRO Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):557-566. doi: 10.1001/jama.2017.9938. PMID 28787506